CLINICAL TRIAL: NCT04749355
Title: A Phase 2, Open-Label, Single Arm, Multi-Center Study to Assess the Efficacy and Safety of BST-236 as a Single Agent in Adults Unfit for Intensive Chemotherapy With Relapsed or Refractory AML or Higher-Risk Myelodysplastic Syndromes
Brief Title: Phase 2, Open-Label, Single Arm Study, With BST-236 in Adults With R/R AML or Higher-Risk MDS
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: BioSight Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BST004
Record Dates: First submitted 2021-02-07; First posted 2021-02-11 (Actual); Last update posted 2023-03-09 (Actual); Status verified 2022-07

CONDITIONS: AML, Adult; MDS; Relapse/Recurrence; Refractory Acute Myeloid Leukemia
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Recurrence

STUDY DESIGN:
Intervention Model Description: Open-label, multi-center, single arm, single agent study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- BST-236 (Experimental): BST-236 Intravenous, 4.5 g/m^2/d or 2.3 g/m^2/d, for 6 days
  Interventions: Drug: BST-236

INTERVENTIONS:
Drug: BST-236 — BST-236 is a conjugate of cytarabine and asparagine, provided as a sterile lyophilized powder for IV administration
  Other Names: Aspacytarabine

SUMMARY:
An open label multi center study to assess the safety and efficacy of BST-236 as single agent in adult patients unfit for standard therapy with Acute Myeloid Leukemia (AML) or higher-risk (HR) Myelodysplastic Syndromes (MDS) who fail to respond or relapsed following first line therapy.

Approximately 20 adult patients with relapsed and/or refractory AML and approximately 20 adult patients with relapsed and/or refractory HR MDS, will be enrolled into the study.

Patients will be treated with 1-2 induction courses and 2-4 maintenance courses. All patients will be followed for 1 year in the study and additional 1 year post study follow-up.

ELIGIBILITY:
1. Documented diagnosis of MDS, according to World Health Organization (WHO) classification and Revised International Prognostic Scoring System (IPSS-R) overall score ≥ 4.5 Or

   Diagnosed AML according to the 2016 revision to the WHO classification of myeloid neoplasms and acute leukemia: ≥20% blasts in peripheral blood or bone marrow
2. Adult ≥18 years of age
3. MDS relapse following treatment with azacitidine or decitabine Or

   MDS failure to achieve complete or partial response or stable disease with hematologic improvement after at least 4 cycles of azacitidine or decitabine, all within the last 1 year Or

   MDS progression while on azacitidine or decitabine treatment irrespective of the number of cycles the patient has received Or

   AML relapse after initial CR/CRi/CRh following treatment with: azacitidine, decitabine, Low-Dose Ara-C (LDAC) , venetoclax+HMA, or venetoclax+LDAC Or

   AML failure to achieve CR, CRh or CRi following at least 4 cycles of azacitidine or decitabine or 2 cycles of venetoclax+HMA or venetoclax+LDAC within the last 1 year.

   Or

   AML progression while on azacitidine, decitabine, LDAC, venetoclax+HMA, venetoclax+LDAC, irrespective of the number of cycles the patient has received.
4. Not able to receive an allogeneic bone marrow transplantation (BMT) at the time of study enrolment.
5. Not eligible for intensive chemotherapy;

   1. Age ≥75 years Or
   2. Age ≥18 years with at least one of the following comorbidities:
   3. Significant heart or lung comorbidities, as reflected by at least one of the following:
   4. Left ventricular ejection fraction (LVEF) ≤50%
   5. Lung diffusing capacity for carbon monoxide (DLCO) ≤65% of expected
   6. Forced expiratory volume in 1 second (FEV1) ≤65% of expected
   7. Chronic stable angina or congestive heart failure controlled with medication
   8. Other comorbidity or conditions that the Investigator judges as incompatible with intensive chemotherapy, which must be documented
   9. ECOG=2
6. Creatinine clearance (estimated by the Modification of Diet in Renal Disease (MDRD) equation or measured by 24 hours urine collection) ≥45 mL/min
7. Liver enzymes (aspartate aminotransferase (AST) and/or alanine aminotransferase (ALT) ≤2.5 times the upper limits of normal (ULN), unless attributed to leukemia (in AML patients)
8. Total bilirubin ≤3 XULN unless due to Gilbert disease
9. Eastern Cooperative Oncology Group (ECOG) performance status ≤ 2
10. Women of reproductive potential must have a negative serum pregnancy test within 48 hours prior to the first day of any BST-236 treatment course
11. Women of reproductive potential must use two forms of effective birth control methods starting from at least 1 month prior to BST-236 first dose and until 3 months following the last BST-236 administration day (acceptable methods of birth control in this study include: surgical sterilization, intrauterine devices, oral contraceptives, contraceptive patch, long-acting injectable contraceptives, or double-barrier method condom or diaphragm with spermicide)
12. Male subjects must agree to refrain from unprotected sex and sperm donation from initial study drug administration until 3 months following the last dose of study drug
13. Subject must voluntarily sign and date an informed consent, approved by an Independent Ethics Committee (IEC)/Institutional Review Board (IRB), prior to the initiation of any screening or study-specific procedures
14. Patient must be able to adhere to the study visit schedule and other protocol requirements

Exclusion Criteria:

1. MDS or AML evolving from a pre-existing myeloproliferative neoplasm (MPN)
2. MDS/MPN including chronic myelomonocytic leukemia (CMML), atypical chronic myeloid leukemia (CML), juvenile myelomonocytic leukemia (JMML) and unclassifiable MDS/MPN
3. Acute promyelocytic leukemia
4. Previous treatment for AML or MDS with drugs other than HMA or LDAC or combinations of venetoclax with either HMA or LDAC
5. Previous allogeneic hematopoietic stem cell transplantation (HSCT) or solid organ transplantation
6. Participation in a previous clinical trial involving use of an investigational drug within 30 days or at least 5 half-lives of tested drug (whichever is shorter) of study day 1
7. Peripheral White Blood Cell (WBC) count >30,000 /µL in the 48 hours prior to first BST-236 dose administration. Hydroxyurea administration or leukapheresis is permitted to meet this criterion
8. Administration of HMA, LDAC, or venetoclax within 14 days prior to Study Day 1
9. Previous treatment with cytarabine at a dose higher than 20 mg/ m2/d
10. Uncontrolled systemic fungal, bacterial, or viral infection (defined as ongoing signs/symptoms related to the infection without improvement despite appropriate antibiotics or other treatment)
11. Any medical or surgical condition, presence of laboratory abnormalities or psychiatric illness that may preclude safe and complete study participation based on the Investigator's judgment
12. Diagnosis of malignant disease (other than AML) within the previous 12 months (excluding basal cell carcinoma of the skin without complications, "in-situ" carcinoma, or other local malignancy excised or irradiated with a high probability of cure and not treated with systemic or topical chemotherapy)
13. Surgical procedure, excluding central venous catheter placement or other minor procedures (e.g. skin biopsy) in the 14 days prior to first BST-236 dose administration
14. History of allergic reactions attributed to compounds of similar chemical composition as BST-236 and/or cytarabine
15. Life expectancy shorter than 3 months attributed to any known medical condition other than AML/MDS
16. In 12 leads ECG, corrected QT interval (QTc)>480msec or history of QT prolongation or Torsades de pointes

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2021-11-14 (Actual); Primary Completion 2023-12-14 (Estimated); Study Completion 2024-03-14 (Estimated)

PRIMARY OUTCOMES:
CR rate | To be assessed 5 months after the last patient was enrolled to the study
  In AML patients -The proportion of patients who achieve a CR per the IWG 2006 Criteria
Overall response rate (ORR) | To be assessed 5 months after the last patient was enrolled to the study
  In MDS patients -Overall response rate (ORR), defined as the proportion of patients who achieve a CR or PR per proposal for modification of the International Working Group (IWG) criteria for MDS, 2006

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - Ochsner LSU Health Shreveport - Academic Medical Center, Shreveport, Louisiana
  - The University of Texas MD Anderson Cancer center, Houston, Texas
  - University of Virginia Cancer Center, Charlottesville, Virginia
  - Seattle Cancer Care Alliance, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No